CLINICAL TRIAL: NCT05018182
Title: To Observe the Pathological Remission Rate and Safety of FOLFOXIRI for Neoadjuvant Treatment of High-risk Locally Advanced Colorectal Cancer With a Single-arm, Open, Prospective Phase II Exploratory Clinical Study
Brief Title: FOLFOXIRI for Neoadjuvant Treatment of High-risk Locally Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meng Qiu, Clinical Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-010
Record Dates: First submitted 2021-08-03; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: High-risk Locally Advanced Colorectal Cancer; Neoadjuvant Chemotherapy; FOLFOXIRI Regimen
MeSH Terms: interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant chemotherapy (Experimental): 4 cycles of neoadjuvant chemotherapy with FOLFOXIRI + operation + 5 cycles of adjuvant chemotherapy with XELOX
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Folinic Acid; Drug: 5FU; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 85 mg/m² Q2w(2 h) before surgery rection and 130 mg/m² Q3w (2 h) after surgery
  Other Names: Eloxatin
Drug: Irinotecan — Irinotecan 150 mg/m² ivgtt(1.5 h) Q2w before surgery rection
  Other Names: Campto
Drug: Folinic Acid — Folinic acid 400 mg/m² ivgtt(2 h) Q2w before surgery rection
  Other Names: Leukovorin
Drug: 5FU — 5-FU 2800 mg/m² civ(46 h) Q2w before surgery rection
  Other Names: 5-Fluorouracil
Drug: Capecitabine — Capecitabine 1000mg/m² d1-14 po Q3w after surgery rection
  Other Names: Xeloda

SUMMARY:
The main cause of recurrence after surgical treatment of colorectal cancer is distant metastasis. Neoadjuvant chemotherapy has potential benefits of improving the effectiveness of chemotherapy. Preoperative chemotherapy may eradicate microscopic metastatic cancer cells earlier than adjuvant chemotherapy, reduce cancer cell spillage during surgery, and lessen the invasiveness of surgical resection. The FOLFOXIRI regimen has been shown to have a high objective efficiency in advanced colorectal cancer. This phase II trial is to explore the pathological remission rate and safety of stage II/III locally advanced colon cancer with high risk of recurrence to FOLFOXIRI regimen of neoadjuvant chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old; Sex: Male or female;
* WHO performance status of 0, 1 or 2
* Histologically proven colorectal carcinoma (defined as cancer that is located >10 cm from the anal verge by endoscopy)
* Unequivocal radiological evidence of locally advanced cancer based on thin slice spiral CT [defined as T4a/b or (and) N2 / fused lymph nodes or (and) positive extramural vascular invasion (EMVI +) or (and) circumferential resection margin (CRM) ≤ 2mm].
* No distant metastases (distant organ or (and) distant lymph node metastases) assessed by CT scan or other radiographic examination.
* For patients with T4b, R0 resection was expected to be achieved, including the necessary combined organ resection，by MDT discussion.
* No history of 5-Fu and platinum drug allergy.
* Adequate bone marrow function: Hb>9g/dl; PLT >100 x 10^9/l; WBC >3.5 x 10^9/l and ANC ≥1.5x10^9/l.
* Adequate hepatobiliary function: ASAT (aspartate aminotransferase) and ALAT (alanine aminotransferase) of 2.5 x ULN (upper limits of normal) or less, Alkaline phosphatase of 2.5 x ULN or less, total bilirubin 1.5 x upper normal level or less.
* Adequate renal biochemistry: GFR >50 ml/min calculated by the Wright or Cockroft formula or EDTA clearance >70 ml/min.
* For female and of childbearing potential, patient must have a negative pregnancy test ≤72hours prior to initiating study treatment and agree to avoid pregnancy during and for 6 months after study treatment. For male with a partner of childbearing potential, patient must agree to use adequate, medically approved, contraceptive precautions during and for 90 days after the last dose of study treatment
* Patient able and willing to provide written informed consent for the study.

Exclusion Criteria:

* Patients with lynch syndrome
* Rectal cancer located 10 cm or less from the anal verge.
* Any patient for whom radiotherapy is advised by the MDT.
* Patient with evidence of distant metastases or peritoneal nodules (M1).
* Severe intestinal complications on initial clinical or imaging assessment: perforation, obstruction, uncontrollable bleeding.
* Another serious medical condition judged to compromise ability to tolerate neoadjuvant therapy and/or surgery.
* Pre-existing or concurrent other malignancies (including concurrent colon cancer), except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix.
* Pregnant or breastfeeding women.
* Patients with severe cardiovascular disease and diabetes mellitus that cannot be easily controlled.
* Persons with mental disorders.
* Patients with severe infections.
* Patients on thrombolytic/anticoagulant therapy, bleeding quality or coagulation disorders; or aneurysms, strokes, transient ischemic attacks, arteriovenous malformations in the past year.
* Previous history of renal disease with urine protein on urinalysis or clinically significant renal function abnormalities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-08-02 (Estimated)

PRIMARY OUTCOMES:
Pathological response | up to 24 weeks
  The rate of Tumor Regression Grade 0-1 in the resected tumour tissue

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 weeks
  Rate of patients with partial or complete response according to modified RECIST criteria.
Pathologic Complete Response (PCR) | up to 24 weeks
  Rate of pathological complete response in the resected tumour tissue
R0 resection rate | up to 24 weeks
  Resection rate, defined as patients with microscopically complete (R0) resection (ITT- population)
Progression Free Survival (PFS) | up to 3 years
  Progression free survival (Medium, Kaplan-Meier-estimation, ITT- population)
Distant metastasis-free survival Metastasis-free survival | up to 3 years
  distant Distant metastasis-free survival (Medium, Kaplan-Meier-estimation, ITT- population)
Overall survival | up to 3 years
  Overall survival (Kaplan-Meier-estimation, ITT- population)
Toxicity and Compliance to study treatment | up to 1 years
  Toxicity according to NCI-CTC criteria v. 4.0 Perioperative toxicity according to Clavien
Molecular markers | up to 1 years
  Evaluation of molecular predictive markers for response and toxicity
Quality of Life to study treatment | up to 1 years
  scores of Quality of Life Questionare-Core 30 of the European Organization for Research and Treatment of Cancer
Number of patients with 30-day post-operative mortality | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Leng, Ph.D, Principal Investigator — Sichuan University
Locations (1):
- Sichuan University West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Leng W, Zhou Y, Yu Y, Meng W, Cao P, Wang Z, Qiu M. Pathological response and safety of FOLFOXIRI for neoadjuvant treatment of high-risk relapsed locally advanced colon cancer: study protocol for a single-arm, open-label phase II trial. BMJ Open. 2023 Jan 31;13(1):e062659. doi: 10.1136/bmjopen-2022-062659. PMID 36720570